CLINICAL TRIAL: NCT00774345
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of Lenalidomide (Revlimid®) as Maintenance Therapy for Patients With B-Cell Chronic Lymphocytic Leukemia Following Second-Line Therapy (The Continuum Trial)
Brief Title: A Study to Evaluate the Efficacy and Safety of Lenalidomide as Maintenance Therapy for Patients With B-Cell Chronic Lymphocytic Leukemia (CLL) Following Second Line Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-CLL-002
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: 1 (Experimental): Lenalidomide po qd on days 1-28 of a 28 day cycle
  Interventions: Drug: Lenalidomide
- Placebo Comparator: 2 (Placebo Comparator): Placebo capsules given orally on days 1-28 of a 28 day cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide capsules given orally on days 1-28 of a 28 day cycle
  Other Names: Revlimid
  Arms: Experimental: 1
Drug: Placebo — Placebo capsules given orally on days 1 - 28 of a 28 day cycle
  Arms: Placebo Comparator: 2

SUMMARY:
The purpose of this study is to determine if lenalidomide (Revlimid®) is safe and effective as a maintenance therapy at improving further the quality of the response you achieved with your last therapy and at prolonging the duration of your response. This study will compare the effects (good and bad) of lenalidomide with the dummy drug.

DETAILED DESCRIPTION:
This is a phase 3, randomized (computer assigned by chance to treatment arm), study being completed an multiple sites to compare the safety and efficacy (how well a drug works) of lenalidomide maintenance therapy to placebo (dummy capsule that contains no lenalidomide or active substances) maintenance therapy.

Patients are assigned by a computer with a 50/50 chance to receive placebo or lenalidomide study treatment. Study drug will be taken once each day until the patient discontinues the study. Patients will remain on study drug until progression of disease.

Patients will visit their study doctor every 28 days until disease progression to complete safety and efficacy assessments. Quality of life assessments will be completed every other month. If a patient who discontinue study drug prior to disease progression (i.e. due to an adverse reaction to the study drug), they will continue to visit the study doctor each month to complete the efficacy assessments up to progression of disease. Safety assessments may include laboratory blood tests, ECG tests and questions about any medical conditions or side effects experienced during the study. Efficacy assessments may include laboratory blood tests and focused physical exams.

Computed tomography (CT) scans along with blood tests and bone marrow samples will be collected to confirm if a patient has improvement of response while on study.

After disease progression, patients will be contacted every 12 weeks for survival information, next CLL treatments and quality of life questions.

Subjects currently on lenalidomide treatment will discontinue lenalidomide treatment immediately and complete the Treatment Discontinuation assessment. The subjects will then transition to the survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Must be greater than or equal to 18 years at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Must have a documented diagnosis of B-cell CLL (IWCLL guidelines for the diagnosis and treatment of chronic lymphocytic leukemia [Hallek, 2008]).
5. Must have been treated with one of the following in first and/or second line:

   * a purine analog-containing regimen
   * a bendamustine-containing regimen
   * an anti-CD20 antibody-containing regimen
   * a chlorambucil-containing regimen
   * an alemtuzumab-containing regimen (for those subjects with a 17p deletion)
6. Must have achieved a minimum response of partial response (PR, nPR, CRi, CR, and MRD-negative CR) (IWCLL guidelines for the diagnosis and treatment of chronic lymphocytic leukemia [Hallek, 2008]) following completion of second-line induction therapy prior to randomization (documentation of response status must be available). Second-line induction therapy must be documented to have been of sufficient duration.
7. Must have completed last cycle of second-line induction no less than 8 weeks (56 days) and no greater than 20 weeks (140 days) prior to randomization.
8. Must have an ECOG performance status score of less than or equal to 2.
9. Females of childbearing potential (FCBP)† must:

   * Have two negative medically supervised pregnancy tests prior to starting of study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices complete and continued sexual abstinence.
   * Either commit to continued abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
10. Male subjects must:

    * Commit to continued abstinence from heterosexual contact or agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after cessation of study therapy.
    * Agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
11. All subjects must:

    * Have an understanding that the study drug could have a potential teratogenic risk.
    * Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy. • Agree not to share study medication with another person.
    * All subjects must be counseled about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Active infections requiring systemic antibiotics.
3. Systemic infection that has not resolved > 2 months prior to initiating lenalidomide treatment in spite of adequate anti-infective therapy
4. Autologous or allogeneic bone marrow transplant as second-line therapy.
5. Pregnant or lactating females.
6. Systemic treatment for B-cell CLL in the interval between completing the last cycle of second-line induction therapy and randomization.
7. Participation in any clinical study or having taken any investigational therapy for a disease other than CLL within 28 days prior to initiating maintenance therapy.
8. Known presence of alcohol and/or drug abuse.
9. Central nervous system involvement as documented by spinal fluid cytology or imaging. Subjects who have signs or symptoms suggestive of leukemic meningitis or a history of leukemic meningitis must have a lumbar puncture procedure performed within two weeks prior to randomization.
10. Prior history of malignancies, other than CLL, unless the subject has been free of the disease for ≥5 years. Exceptions include the following:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
11. History of renal failure requiring dialysis.
12. Known Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), and/or active Hepatitis C Virus (HCV) infection.
13. Prior therapy with lenalidomide.
14. Evidence of TLS per the Cairo-Bishop definition of laboratory TLS (subjects may be enrolled upon correction of electrolyte abnormalities).
15. Any of the following laboratory abnormalities:

    * Calculated (method of Cockroft-Gault) creatinine clearance <60 mL/min.
    * Absolute neutrophil count (ANC) <1,000/μL (1.0 X 109/L)
    * Platelet count <50,000/μL (50 X 109/L)
    * Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 3.0 x upper limit of normal (ULN)
    * Serum total bilirubin >2.0 mg/dL (with the exception of Gilbert's Syndrome)
16. Grade 4 rash due to prior thalidomide treatment
17. Uncontrolled hyperthyroidism or hypothyroidism
18. Venous thromboembolism within one year
19. Greater than or equal to Grade-2 neuropathy
20. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
21. Disease transformation (active) (ie, Richter's Syndrome, prolymphocytic leukemia)
22. Known allergy to allopurinol for subjects assessed with PR following their second-line induction therapy.
23. Prisoners.
24. More than 2 prior lines of CLL therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2009-01-27 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Delarue, MD, Study Director — Celgene Corporation
Locations (241):
- United States (56):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Pacific Coast Hematology Oncology, Fountain Valley, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University Stanford, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Pasco Hernando Oncology Associates, PA, Brooksville, Florida
  - Memorial Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialist, Tavares, Florida
  - Florida Hospital Cancer Institute Waterman, Tavares, Florida
  - Augusta Oncology Associates, P.C., Augusta, Georgia
  - Northwest Georgia Oncology Centers, PCWilliam S. Gibbons Center Research Institute, Marietta, Georgia
  - Northwestern University, Division of Hematology Oncology, Dept. of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Hematology Oncology Assoc. of IL Orchard Research LLC, Skokie, Illinois
  - Floyd Memorial Cancer Center of Indiana, a division of Floyd Memorial Hospital and Health Services, New Albany, Indiana
  - McFarland Clinic, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Ochsner Medical Institutions, New Orleans, Louisiana
  - Clinical Unit for Research Trials in Skin CURTIS Massachusetts General Hospital, Boston, Massachusetts
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - The Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Biomedical Research Alliance of New York, LLC, New Hyde Park, New York
  - SUNY Upstate Medical University Medicine Oncology, Syracuse, New York
  - Westchester County Medical Center, Valhalla, New York
  - Wake Forest Univ. Health Sciences Outpatient Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Gabrail Cancer Center Research, Dover, Ohio
  - Trilogy Cancer Care, Wooster, Ohio
  - Kaiser Permanente Northwest Oncology Hematology, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Drexel University, College of Medicine, Clinical Research Group, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Abington Hematology Oncology Associates Inc, Willow Grove, Pennsylvania
  - Charleston Hematology Oncology P.A., Charleston, South Carolina
  - M. Francisco Gonzalez, MD, PA, Sumter, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Gundersen Clinic Lutheran Hospital, La Crosse, Wisconsin
- Australia (13):
  - Concord Hospital, Concord, New South Wales
  - Haematology and Oncology Clinics of Australasia, South Brisbane, Queensland
  - IMVS, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park
  - Royal Prince Alfred Hospital, Camperdown
  - Peter MacCallum Cancer Centre, East Melbourne
  - Frankston Hospital, Farkston
  - St. Vincent Hospital, Fitzroy
  - Nepean Hospital, Kingswood, NSW
  - Clinical Trials Unit The St George Hospital, Kogarah
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal North Shore HospitalDepartment of HematologyLevel 4, St Leonards
  - The Queen Elizabeth Hospital, Woodville
- Austria (3):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Hospital Bamherzige Schwestern, Linz
  - Medical University of Vienna Internalmedicine 1, Hematology, Vienna
- Belgium (8):
  - AZ Sint-Jan AV Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - UZ Gent Hematology, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU Mont -Godinne, Yvoir
- Canada (8):
  - Regional Health Authority B-Saint John Regional Hospital, Saint John, New Brunswick
  - General Hospital, Eastern Health, St. John's, Newfoundland and Labrador
  - CDHA Centre for Clinical Research, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CIUSSS de l'Est-de-l'Ile-de-Montreal, Montreal/Quebec, Quebec
  - Hopital De L'Enfant-Jesus, Québec
- Oncomedica S.A., Montería, Colombia
- Czechia (6):
  - Interni hematoonkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Poliklinika Agel Novy Jicin, Nový Jičín
  - Faculty Hospital Plzen, Pilsen
  - Faculty Hospital Kralovske Vinohrady, Prague
  - General Faculty Hosital1.Internal Clinic, Prague
- Denmark (3):
  - Rigshospitalet University Hospital, Copenhagen
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- France (12):
  - Hopital Aviecenne, Bobigny
  - Bergonie Institut, Bordeaux
  - CMRU-Hotel Dieu Service Hematologie Clinique et Therapie Cellulaire, Clermont-Ferrand
  - CHU Hopital Michallon, Grenoble
  - Centre Hospitalier Lyon Sud, Lyon
  - Cetre Hospitalier Hotel-Dieu, Nantes
  - Hopital de l'Archet 1, Nice
  - Hopital Petie- SalpetriereDepartment d'Hematologie, Paris
  - CHU La Miletrie, Poitiers
  - CHU de Reims, Reims
  - CLCC H BecquerelHematology, Rouen
  - Hopital Bretonneau, Tours
- Germany (13):
  - Charite, Campus Benjamin Franklin, Medizinische Klinik III, Berlin
  - Klinikum der Universitat zu Koln, Cologne
  - Universitaetsklinikum EssenZentrum fuer Innere Medizin, Essen
  - Innere Medizin Klinikum Frankfurt Oder GmBH, Frankfurt (Oder)
  - Universitaetsklinikum FreiburgInnere Med.1, Haematologie, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Praxis fuer Haematologie und Onkologie Koblenz, Koblenz
  - Universitatsklinikum Leipzig, Leipzig
  - Mannheimer Onkologie Praxis, Mannheim
  - Stadtisches Klinikum Munchen GmbH, München
  - TU München - Klinikum rechts der Isar, München
  - Facharzte fur Innere Medizin Hämatologie und Onkologie Gemeinschaftspraxis, Münster
  - University Hospital of Ulm, Ulm
- Hungary (7):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Petz Aladar Country Hospital, Győr
  - Kaposi Mor Oktato Korhaz, Kaposvár
  - Pecsi Tudomanyegytem Altalanos Orvostudomanyi Kar, Pécs
  - Szegedi TudomanyegyetemII Belgyogyaszati Klinika, Szeged
  - Komarom-Esztergom Megye Onkormanyzat Szent Borbala Korhaza, Tatabánya
- Ireland (2):
  - St James's Hospital, Dublin
  - Midwestern Regional Hospital, Limerick
- Israel (12):
  - Ha'Emek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Bnei Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (25):
  - Azienda Ospedaliera Poloclinico di Bari, Bari
  - Istituto dei Tumori Giovanni Paolo II di Bari, Bari
  - AO Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Vittorio Emanuele-Ferrarotto, Catania
  - A.O. Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliera Annunziala, Cosenza
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria OORR Foggia, Foggia
  - Azienda Ospedaliera San Martino, Genova
  - IRCSS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Istituto Oncologico Europeo, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Ospedale Cardarelli, Naples
  - Policlinico Universitario Federico II, Naples
  - Universita del Piemonte Orientale, Novara
  - Universita degli Studi di Padova, Padua
  - Azienda Ospedaliera Ospedale San Carlo, Potenza
  - Ospedale Sant'Eugenio, Rome
  - Azienda Policlinico Umberto I, Universita La Sapienzadi Roma, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - Osp. S.Giovanni Battista Le Molinette, Torino
  - Ospedale Umberto I, Torrette Di Ancona
  - Ospedale San Bortolo di Vicenza, Vicenza
- Instituto Biomedico de Investigacion AC, Aguascalientes, Mexico
- VU University Medical Center, Amsterdam, Netherlands
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Middlemore Clinical Trials, Manukau
  - North Shore Hospital, Takapuna
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Specjalistyczny Szpital miejski im. Kopernika, Torun
  - Centralny Szpital Kliniczny MON, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Portugal (3):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Dia de Hematologia, Lisbon
  - Instituto Portugues Oncologia do Porto Francisco Gentil EPE, Porto
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf Spiridon Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (17):
  - Archangelsk Regional Clinical Hospital, Arkhangelsk
  - City Hospital 8, Barnaul
  - GMU Republic clinical hospital, Kazan'
  - Krasnoyarsk Regional Clinical Hospital, Krasnoyarsk
  - Institution of Russian Academy of Medical Sciences Russian Oncological Research Centre n.a. N. N. Bl, Moscow
  - State Budgetary Institution of the City of Moscow, Moscow
  - NUZ Central Clinical Hospital, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - MUZ City Clinical Hospital 2, Novosibirsk
  - Federal State Budgetary Establishment Medical Radiological Research Center Ministry of Health and so, Obninsk
  - FGU Russian Scientific Research Institute of Haematology and Transfusiology of Federal Agency, Saint Petersburg
  - GUS Leningrad Regional Clinical Hospital, Saint Petersburg
  - St. Petersburg Pavlov State Medical Univ, Saint Petersburg
  - Federal State Institution Federal Centre of Heart, Blood and Endocrinology of Rosmedtechnologies, Saint Petersburg
  - Saratov State Medical University, Saratov
  - GUZ Volgograd Regional Clinical Oncology, Volgograd
  - State Healthcare Institution Sverdlovsk regional clinical hospital 1, Yekaterinburg
- South Africa (5):
  - Groote Schuur Hospital, Cape Town
  - University Witwatersrand Oncology, Parktown
  - Pretoria Academic Hospital, Pretoria
  - Mary Potter Oncology Centre, Pretoria
  - Wilgers Oncology CentreWilgrers Hospital, Pretoria
- Spain (14):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall D hebron, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda
  - Virgen de la Victoria Hospital Malaga, Málaga
  - Hospital General Universitario Morales Messeguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario, Valencia
- Sweden (3):
  - Skane University Hospital, Lund
  - Stockholm South Hospital, Stockholm
  - Karolinska University, Stockholm
- United Kingdom (14):
  - Royal Bournemouth General Hospital, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Gartnavel General Hospital, Glasgow
  - John Radcliffe Hospital, Headington
  - Saint James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - St. Bartholomew's and The Royal London Hospital, London
  - Guy's and St. Thomas' Hospital, London
  - King's College Hospital, London
  - St George's Healthcare NHS Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Singleton Hospital, Southwest Wales Cancer Inst, Swansea
  - Sandwell Hospital, West Bromwich

REFERENCES:
- [Derived] Chanan-Khan AA, Zaritskey A, Egyed M, Vokurka S, Semochkin S, Schuh A, Kassis J, Simpson D, Zhang J, Purse B, Foa R. Lenalidomide maintenance therapy in previously treated chronic lymphocytic leukaemia (CONTINUUM): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Haematol. 2017 Nov;4(11):e534-e543. doi: 10.1016/S2352-3026(17)30168-0. Epub 2017 Sep 25. PMID 28958469

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 317 randomized and 315 treated.
Groups:
- Lenalidomide; Placebo: 2.5mg QD PO with escalation after 28 days to 5mg QD PO x 28 days, only if the 2.5mg dose was tolerated. Participants could be escalated to 10mg QD PO x 28 days, but only after 5 continuous cycles at 5mg and only if 5mg was well tolerated and if those participants had not achieved MRD-negative CR
Period: Pre-treatment
Arm/Group | Lenalidomide | Placebo
Started (Started = Randomized) | 160 | 157
Completed (Completed = Treated) | 158 | 157
Not Completed | 2 | 0
Not completed — Other reasons | 2 | 0
Period: Treatment
Arm/Group | Lenalidomide | Placebo
Started | 158 | 157
Participants Escalated to 5mg | 129 | 149
Participants Escalated to 10mg | 68 | 88
Completed | 0 | 0
Not Completed | 158 | 157
Not completed — Adverse Event | 61 | 15
Not completed — Progressive Disease without histologic transformation | 51 | 111
Not completed — Progressive Disease with histologic transformation | 4 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 4 | 0
Not completed — Other Reasons | 32 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Placebo | Total
Number analyzed (Participants) | 160 | 157 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (8.08) | 62.5 (8.85) | 62.7 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 115 | 113 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 153 | 156 | 309
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 154 | 150 | 304
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from randomization to death from any cause. OS will be censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: Up to approximately 11 years
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 160 | 157
Months | 95.09 [70.35 to 103.52] | 73.28 [59.98 to 102.98]
Statistical Analysis 1: Comparison: Lenalidomide vs Placebo; Test type: Superiority; p = 0.276, Log Rank — The p-value is based on a stratified log-rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.15] — Based on the stratified cox proportional hazards model comparing the hazard functions associated with the treatment groups

2. Secondary Outcome: Progression Free Survival 2 (PFS2)
Description: Progression Free Survival (PFS2) assessed by investigator is defined as the time from randomization to the second objective disease progression, or death from any cause, whichever occurs first.
Time Frame: Up to 6 years
Population: All randomized evaluable participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 160 | 154
Months | NA [49.5 to NA] — Median and Upper Limit not reached because of too few events to evaluate | 35.9 [27.4 to NA] — Too few events to estimate the upper limit of the confidence interval

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with adverse events (AEs) that measure type, frequency and severity of AEs graded by National Cancer Institute Common Terminology Criteria (NCI CTCAE V 3.0) including any grade adverse events (AEs), Grade 3-4 AEs, AEs related to study drug, grade 3-4 AEs related to study drug.
Time Frame: From first dose to 30 days post last dose (up to 9 years)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 158 | 157
Participants
  Adverse Events (AEs) | 155 | 149
  Grade 3-4 AEs | 136 | 73
  AEs related to Study drugs | 143 | 98
  Grade 3-4 AEs related to Study drugs | 117 | 41

ADVERSE EVENTS:
Time Frame: Up to 9 years
Arm/Group | Lenalidomide | Placebo
All-Cause Mortality (participants affected / at risk) | 78/158 | 80/157
Serious Adverse Events (participants affected / at risk) | 99/158 | 49/157
Other Adverse Events (participants affected / at risk) | 152/158 | 140/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=158) | Placebo (N=157)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 3 | 2
Autoimmune pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 49 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0
Optic neuropathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Soft tissue inflammation (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bone tuberculosis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lymph node abscess (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 7 | 8
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Sinusitis bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viral labyrinthitis (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Blood bicarbonate decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Demyelination (Nervous system disorders) | 1 | 0
Diplegia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=158) | Placebo (N=157)
Anaemia (Blood and lymphatic system disorders) | 9 | 7
Leukopenia (Blood and lymphatic system disorders) | 12 | 2
Neutropenia (Blood and lymphatic system disorders) | 106 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 19
Abdominal pain (Gastrointestinal disorders) | 18 | 9
Abdominal pain upper (Gastrointestinal disorders) | 9 | 4
Constipation (Gastrointestinal disorders) | 27 | 8
Diarrhoea (Gastrointestinal disorders) | 65 | 26
Dyspepsia (Gastrointestinal disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 26 | 27
Vomiting (Gastrointestinal disorders) | 12 | 13
Asthenia (General disorders) | 10 | 2
Chills (General disorders) | 10 | 1
Fatigue (General disorders) | 56 | 54
Influenza like illness (General disorders) | 11 | 2
Oedema peripheral (General disorders) | 16 | 12
Pyrexia (General disorders) | 28 | 17
Bronchitis (Infections and infestations) | 22 | 12
Herpes zoster (Infections and infestations) | 9 | 9
Influenza (Infections and infestations) | 14 | 3
Lower respiratory tract infection (Infections and infestations) | 12 | 7
Nasopharyngitis (Infections and infestations) | 16 | 18
Oral herpes (Infections and infestations) | 10 | 7
Pharyngitis (Infections and infestations) | 10 | 7
Pneumonia (Infections and infestations) | 10 | 2
Respiratory tract infection (Infections and infestations) | 14 | 10
Sinusitis (Infections and infestations) | 16 | 5
Upper respiratory tract infection (Infections and infestations) | 31 | 28
Viral infection (Infections and infestations) | 8 | 5
Blood bilirubin increased (Investigations) | 8 | 4
Weight decreased (Investigations) | 22 | 14
Weight increased (Investigations) | 5 | 9
Decreased appetite (Metabolism and nutrition disorders) | 15 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 6
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 9
Dizziness (Nervous system disorders) | 16 | 9
Headache (Nervous system disorders) | 17 | 14
Insomnia (Psychiatric disorders) | 10 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 10 | 3
Erythema (Skin and subcutaneous tissue disorders) | 8 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 30 | 31
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 9
Rash (Skin and subcutaneous tissue disorders) | 42 | 13
Hypertension (Vascular disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT00774345/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT00774345/SAP_001.pdf